CLINICAL TRIAL: NCT02153749
Title: Regulation of Craving: Brief Neurocognitive Training and Neural Mechanisms
Brief Title: Effects of Brief Training on Craving Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1210010970; P50DA009241 (NIH)
Record Dates: First submitted 2014-05-23; First posted 2014-06-03 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Nicotine Addiction
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Regulation of Craving (Experimental): Training in craving regulation component of Cognitive Behavioral Therapy(CBT) for addictions.
  Interventions: Behavioral: Cognitive Regulation of Craving
- Mindfulness-Based Regulation of Craving (Experimental): Training in craving regulation component of Mindfulness Based Therapy(MBT) for addiction.
  Interventions: Behavioral: Mindfulness-Based Regulation of Craving
- No training control (No Intervention): No training sessions will be provided in this arm.

INTERVENTIONS:
Behavioral: Cognitive Regulation of Craving — Regulation strategy practice: Participants will be trained to use a CBT-based cognitive regulation strategy. They will be asked to think of their individualized negative consequences for and thing of them when they see the instruction "LATER" during the task. Participants will practice using this strategy for multiple cigarette stimuli. High-Risk Situation Practice: Participants will identify 10 situations in which they usually smoke, or are likely to smoke in the next 48 hours. For each situation, they will be asked to practice using the strategy and to plan to use this strategy to regulate craving in daily life.
  Arms: Cognitive Regulation of Craving
Behavioral: Mindfulness-Based Regulation of Craving — Each training session in this condition will be identical to the CBT-based training session described, with the exception of the strategy being trained. Specifically, participants will be trained in using the MBT-based strategy ("notice craving and accept the feeling without judgment or reaction"). To do so, they will be asked to generate their own non- reactive responses to craving (e.g., "I can just sit here and notice this. I can ask myself, 'can I be ok with this feeling?'") Participants will then be instructed to think of those accepting and non-reactive responses when they see the instruction "ACCEPT" during the task. All other components will be identical.
  Arms: Mindfulness-Based Regulation of Craving

SUMMARY:
The investigators propose that brief training in regulation of craving may increase the efficacy of smoking cessation, but that training in cognitive vs. mindfulness-based strategies may operate via different psychological and neural mechanisms.

DETAILED DESCRIPTION:
The investigators propose to test the efficacy of such training by randomizing 126 cigarette smokers to the following conditions: 1) brief training in cognitive regulation of craving 2) mindfulness-based training, and 3) control or no training. Training will be delivered in 6x1 hour computerized sessions over four weeks. Control subjects simply fill out assessments during their visits. Participants who were randomized into the cognitive or mindfulness training complete Regulation of Craving (ROC) training sessions of approximately 60-90 minutes. If randomized into the cognitive regulation training, subjects will be trained to use a cognitive strategy that instructs them to think of all the negative outcomes associated with continued cigarette smoking. If randomized into the MBT-based regulation training, subjects will be trained to use a mindfulness strategy that instructs them to notice and accept their feelings of craving without judgment or intent to act upon them. After all training sessions are completed, there is a 4 week and 12 week follow-up. The investigators will evaluate the effects of training on craving and regulation of craving measured by self-report and functional magnetic resonance imaging during the Regulation of Craving(ROC) task administered pre- and post- treatment, as well as smoking.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 60
2. Smoking 10 or more cigarettes per day,
3. Score >4 on the Fagerstrom Test For Nicotine Dependence (FTND)
4. Treatment seeking (motivated to quit or reduce smoking; >6 on a 10 point likert scale)
5. Fluent English speaker
6. Can commit to the full length of the protocol (~8 weeks) and
7. Are willing to be randomized to treatment condition.

Exclusion Criteria:

1. Current or past comorbid Axis I disorders (assessed via the Mini Psychiatric Interview Diagnosis; MINI)
2. Current use of any psychoactive medications that have not been at a stable dose for the past 6 months, are used as mood stabilizers, or are used as smoking cessation treatments (e.g. varenicline).
3. Serious or unstable medical condition within past 6 months
4. Use of an investigational drug currently or within past 30 days
5. Use of psychoactive medications or those that affect blood flow
6. Other conditions contra-indicated for MRI (e.g., claustrophobia, presence of ferromagnetic metal in the body, prior head trauma with loss of consciousness, color blindness, hypertension, pregnancy).
7. For females only: pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2015-09; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in Self-report Craving level | Baseline to 4 weeks
  ROC task performance, as change from pre- to post- training in (1) craving (operationalized as self-reported craving on craving trials). (2) strategy-specific regulation (operationalized as scores on regulation trials using the trained strategy: LATER/control trials for CBT-based training, ACCEPT/mindfulness trials for MBT-based training). (3) strategy-non-specific regulation (scores on regulation - using the non-trained strategy: LATER trials for MBT-based training, ACCEPT trials for CBT-based training).
% change in craving and control related neural activity measured via functional magnetic resonance imaging (fMRI). | Baseline to 4 weeks
  The neural activity component will be calculated as change from pre-to post- training during fMRI ROC task, including (1) craving- related activity (operationalized as neural reactivity in "craving regions" including Ventral Striatum, ventral medial Pre-Frontal Cortex); (2) neural substrates of control during regulation of craving (operationalized as neural activity in "control regions" including dorsal lateral and ventral lateral prefrontal cortex).
Change in Smoking | baseline to 4 weeks
  Measurement of reduction in cigarette smoking, measured by self report/cotinine/Carbon dioxide(CO2), and FTND smoking severity

SECONDARY OUTCOMES:
Change in Cognitive Control & Affective Reactivity Behavioral Assessments | baseline to 4 weeks
  Detection of generalized effects of the training on affective reactivity and cognitive control, including: (1) Distress Tolerance, (2) CANTAB neuropsychological assessments, and (3) Drug Risk Response Task (DRRT) to measure regulation skills acquisition.
Change in general neural activity measured via fMRI | Baseline to 4 weeks
  Determination if the effects of training generalize to other measures of cognitive control/distress tolerance, using fMRI task neural activity.

OTHER OUTCOMES:
Gender | 4 weeks
  Whether gender moderates any of the findings

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kober, Ph.D., Principal Investigator — Yale University
Locations (1):
- Clinical & Affective Neuroscience Lab, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Witkiewitz K, Bowen S, Douglas H, Hsu SH. Mindfulness-based relapse prevention for substance craving. Addict Behav. 2013 Feb;38(2):1563-1571. doi: 10.1016/j.addbeh.2012.04.001. Epub 2012 Apr 6. PMID 22534451
- [Background] Ferguson SG, Shiffman S. The relevance and treatment of cue-induced cravings in tobacco dependence. J Subst Abuse Treat. 2009 Apr;36(3):235-43. doi: 10.1016/j.jsat.2008.06.005. Epub 2008 Aug 20. PMID 18715743
- [Background] Elwafi HM, Witkiewitz K, Mallik S, Thornhill TA 4th, Brewer JA. Mindfulness training for smoking cessation: moderation of the relationship between craving and cigarette use. Drug Alcohol Depend. 2013 Jun 1;130(1-3):222-9. doi: 10.1016/j.drugalcdep.2012.11.015. Epub 2012 Dec 21. PMID 23265088
- [Background] Carroll KM. Therapy Manuals for Drug Addiction. A Cognitive-Behavioral Approach: Treating Cocaine ￼Addiction. In: Abuse NIoD, ed. Bethesda, MD: National Institute of Drug Abuse; 1998.
- [Background] Brewer JA, Mallik S, Babuscio TA, Nich C, Johnson HE, Deleone CM, Minnix-Cotton CA, Byrne SA, Kober H, Weinstein AJ, Carroll KM, Rounsaville BJ. Mindfulness training for smoking cessation: results from a randomized controlled trial. Drug Alcohol Depend. 2011 Dec 1;119(1-2):72-80. doi: 10.1016/j.drugalcdep.2011.05.027. Epub 2011 Jul 1. PMID 21723049
- [Background] Kober H, Kross EF, Mischel W, Hart CL, Ochsner KN. Regulation of craving by cognitive strategies in cigarette smokers. Drug Alcohol Depend. 2010 Jan 1;106(1):52-5. doi: 10.1016/j.drugalcdep.2009.07.017. Epub 2009 Sep 11. PMID 19748191
- [Background] Kober H, Mende-Siedlecki P, Kross EF, Weber J, Mischel W, Hart CL, Ochsner KN. Prefrontal-striatal pathway underlies cognitive regulation of craving. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14811-6. doi: 10.1073/pnas.1007779107. Epub 2010 Aug 2. PMID 20679212
- [Background] Westbrook C, Creswell JD, Tabibnia G, Julson E, Kober H, Tindle HA. Mindful attention reduces neural and self-reported cue-induced craving in smokers. Soc Cogn Affect Neurosci. 2013 Jan;8(1):73-84. doi: 10.1093/scan/nsr076. Epub 2011 Nov 22. PMID 22114078
- [Background] Tang YY, Tang R, Posner MI. Brief meditation training induces smoking reduction. Proc Natl Acad Sci U S A. 2013 Aug 20;110(34):13971-5. doi: 10.1073/pnas.1311887110. Epub 2013 Aug 5. PMID 23918376
- [Derived] Roos CR, Harp NR, Vafaie N, Gueorguieva R, Frankforter T, Carroll KM, Kober H. Randomized trial of mindfulness- and reappraisal-based regulation of craving training among daily cigarette smokers. Psychol Addict Behav. 2023 Nov;37(7):829-840. doi: 10.1037/adb0000940. Epub 2023 Aug 3. PMID 37535555